CLINICAL TRIAL: NCT01689454
Title: Prospective Randomized Controlled Trail to Assess the Efficacy of EmbryoGen Culture Medium to Improve Ongoing Pregnancy and Implantation Rates in IVF Treatments of Patients With a Previous History of Implantation Failure
Brief Title: ISM1 Versus EmbrioGen Media for Embryo Culture With Previous Failure Implantation in ART Treatments
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Biogenesi (Other)
Responsible Party: Sponsor
Other Study IDs: EG48BSept12; EG2 (Other: Biogenesi Reproductive Medicine Centre)
Record Dates: First submitted 2012-09-10; First posted 2012-09-21 (Estimated); Last update posted 2012-09-21 (Estimated); Status verified 2012-09

CONDITIONS: Infertility; Implantation Failure
Keywords: IVF; embryo culture; Ongoing pregnancy rate; Ongoing implantation rate; Miscarriage
MeSH Terms: conditions — Infertility; Abortion, Spontaneous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- IVF treatment ISM1: Embryo culture in ISM1 medium
- IVF treatment EG: Embryo culture in EmbryoGen medium

SUMMARY:
Recently, it has been suggested that culture of embryos in EmbryoGen medium can increase the live birth rate in IVF patients with a previous history of pregnancy loss.

Couples requiring IVF treatment and with a past experience of implantation failure will be included in the study.

Controlled ovarian stimulation protocol will consist of an agonist down regulation and follicular stimulation by recombinant FSH. Fertilization will be achieved by standard IVF or intracytoplasmic sperm injection. Fertilized eggs will be cultured in 6% CO2, 5% O2, 89% N2 atmosphere in microdrops. In the treatment group EmbryoGen culture medium (EG, Origio, Måløv, Denmark) will be adopted throughout the culture period. In the control group, inseminated oocytes will be cultured in standard culture conditions, i.e. IMS1 medium (ISM1, Origio, Måløv, Denmark), maintaining unchanged all other culture conditions.

Procedures of embryo transfer, will be carried out on day 2 using EmbryoGen or ISM1 respectively. The endometrial support will be the same in the two groups.

ELIGIBILITY:
Inclusion Criteria:

* women experiencing at least two (maximum 4) failures of implantation after ART treatments (with elective embryo transfer)

Exclusion Criteria:

* Frozen spermatozoa
* Frozen oocytes
* women PCO and PCOS
* women with previous pregnancy, miscarriage or biochemical pregnancy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Infertile couple with an indication for standard IVF or intracytoplasmic sperm injection. Moreover all couples had previous implantation failures after ART treatment (minimun 2 maximun 4 embryo replacements).
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2012-09; Primary Completion 2013-06 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Ongoing Pregnancy Rate after 12 weeks of gestation | 12 weeks after conception

SECONDARY OUTCOMES:
Ongoing Implantation Rate after 12 weeks of gestation | 12 weeks after conception

CONTACTS AND LOCATIONS:
Overall Officials: Mariabeatrice Dal Canto, PhD, Principal Investigator — Biogenesi Reproductive Medicine Centre
Locations (1):
- Biogenesi Reproductive Medicine Centre, Monza, MB, Italy

REFERENCES:
- [Background] Agerholm I, Loft A, Hald F, Lemmen JG, Munding B, Sorensen PD, Ziebe S. Culture of human oocytes with granulocyte-macrophage colony-stimulating factor has no effect on embryonic chromosomal constitution. Reprod Biomed Online. 2010 Apr;20(4):477-84. doi: 10.1016/j.rbmo.2009.12.026. Epub 2009 Dec 28. PMID 20129825